CLINICAL TRIAL: NCT04098679
Title: CONCEPTT Kids Childhood Adiposity and Neurodevelopmental Outcomes Among Offspring of Women With Type 1 Diabetes: A Follow up Study of the CONCEPTT Randomized Control Trial
Brief Title: Childhood Adiposity and Neurodevelopmental Outcomes Among Offspring of Women With Type 1 Diabetes (CONCEPTT Kids)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: SRI International (Industry); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: REB14-2146_MOD2
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Neurologic Disorder; Adiposity
Keywords: Type 1 diabetes; Offspring; Continuous glucose monitoring
MeSH Terms: conditions — Nervous System Diseases; Obesity; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a follow-up study of children born to mothers who participated in the CONCEPTT Trial. CONCEPTT (a multicentre randomized controlled trial of continuous glucose monitoring (CGM) in women with Type 1 diabetes during pregnancy).

The purpose of this study is to examine the association of maternal glycemic measures on childhood intelligence quotient (IQ), behavioural outcomes, language scores and weight measures. The children of the women who participated in CONCEPTT will be assessed.

DETAILED DESCRIPTION:
The assessments will occur between the children's ages of 3-7 years. The assessment will include obtaining consent and child measurements including weight, height, waist circumference and skinfold thickness (at the triceps, subscapular, flank and quadriceps). Body mass index (BMI) and Waist-Height ratio will be calculated.

The other procedures will include:

1. the Wechsler Preschool and Primary Scale of Intelligence-Fourth Edition (1);
2. ADHD Rating Scale IV (2) and ADHD Rating Scale-IV Preschool Version (3);
3. Social Responsiveness Scale-2 for ASD behaviours (4);
4. Children's performance on the Speed Naming and Phonological Processing subscales of the NEPSY-II (5)
5. Parent reported language development on the Children's Communication Checklist-2 for children over four years of age (6) or the Language Use Inventory (LUI) for children 36 to 47 months of age (7).

Basic demographic questions will be asked regarding the child's mother and father including age, ethnicity, education, occupation, family arrangement, presence of major illnesses, and diabetes complications. Questions regarding maternal diabetes, maternal and paternal family history of diabetes and risk factors for heart disease will be collected at the clinic visit.

ELIGIBILITY:
Inclusion Criteria:

* Children of women who participated in the CONCEPTT trial at selected recruiting sites.

Exclusion Criteria:

* Children (of women who participated in the CONCEPTT trial) with major congenital anomalies will be assessed on a case by case basis to determine eligibility.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants, aged 3 to 7 years
Sampling Method: Non-Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
IQ | 2 years
  IQ assessed by the Wechsler Preschool and Primary Scale of Intelligence - Fourth Edition (WPPSI-IV)

SECONDARY OUTCOMES:
ADHD | 2 years
  Attention Deficit Hyperactive Disorder (ADHD) Rating Scale-IV and Attention Deficit Hyperactive Disorder Rating Scale-IV Preschool Version. It is an 18-item questionnaire that requires the respondent to rate the frequency of occurrence of ADHD symptoms. The respondent rates each item on a scale of 0 (not at all) to 3 (very often).
  The scale yields scores for an Inattentive, Hyperactive/Impulsive and Total Scale. The subscales are Inattention Factor and Hyperactive/Impulsive Factor.
ASD | 2 years
  Social Responsiveness Scale-2 questionnaire results for Autism Spectrum Disorder behaviours. It is an 65-item questionnaire that requires the respondent to describe the child's behaviour. The respondent rates each item on a scale of 1 (not true) to 4 (almost always true). The scale yields scores for autism spectrum disorders for total score discussion of social behaviour and social interactions.
NEPSY-II | 2 years
  The NEPSY-II stands for "A Developmental NEuroPSYchological Assessment". Children's language skills assessed using the Speed Naming and Phonological Processing subscales of the NEPSY-II testing results. Phonological Processing is a subtest composed of phonological processing tasks designed to assess phonemic awareness. Speed Naming is a timed subtest designed to assess rapid semantic access to and production of names of colors, shapes, sizes, letters, or numbers.
CCC-2/LUI | 2 years
  Parent reported language development on the Children's Communication Checklist-2 (CCC_2) for children over four years of age or the Language Use Inventory (LUI) for children 36 to 47 months of age questionnaire results. The Children's Communication Checklist - Seconda Edition has 70 Statements that refer to difficulties children may have that affect their ability to communicate. Rating key is 0 (less than once a week or never) to 3 (several times, more than twice, a day, or always). Total score is used.
Demographics | 2 years
  Data form to be completed by parents will ask about their level of education, sex, gender, socioeconomic status, height, and any neurodevelopmental or other medical diagnoses in their enrolled child
Adiposity | 2 years
  Childhood adiposity measures: weight, height, waist circumference and skinfold thickness (at the triceps, subscapular, flank and quadriceps). Body mass index (BMI) and Waist-Height ratio will be calculated using standardized procedures

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Yamamoto, MD MSc FRCPC, Principal Investigator — University of Calgary
Locations (4):
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - Lawson Health Research Institute, London, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
There is no plan for individual level data to be shared with other researchers

REFERENCES:
- [Result] Feig DS, Donovan LE, Corcoy R, Murphy KE, Amiel SA, Hunt KF, Asztalos E, Barrett JFR, Sanchez JJ, de Leiva A, Hod M, Jovanovic L, Keely E, McManus R, Hutton EK, Meek CL, Stewart ZA, Wysocki T, O'Brien R, Ruedy K, Kollman C, Tomlinson G, Murphy HR; CONCEPTT Collaborative Group. Continuous glucose monitoring in pregnant women with type 1 diabetes (CONCEPTT): a multicentre international randomised controlled trial. Lancet. 2017 Nov 25;390(10110):2347-2359. doi: 10.1016/S0140-6736(17)32400-5. Epub 2017 Sep 15. PMID 28923465